CLINICAL TRIAL: NCT01258790
Title: Using Transcranial Magnetic Stimulation to Reduce Tics
Brief Title: Repetitive Transcranial Magnetic Stimulation to Reduce Tics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #: 2010-2689
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Tourette Syndrome
Keywords: TS; tics; tourette
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Repetitive Transcranial Magnetic Stimulation (Sham Comparator): Eight sessions of Repetitive Transcranial Magnetic Stimulation, in the form of Continuous Theta Burst Stimulation, was delivered over the Supplementary Motor Area over 2 days using a Sham TMS coil.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation
- Active Repetitive Transcranial Magnetic Stimulation (Experimental): Eight sessions of Repetitive Transcranial Magnetic Stimulation, Continuous Theta Burst Stimulation, was delivered over the Supplementary Motor Area over 2 days using an Active Magstim Figure-8 TMS coil.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Sham Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (RTMS) is a relatively new technology that allows for targeted noninvasive stimulation of the brain. RTMS is currently FDA-cleared for the treatment of refractory depression. It is also used experimentally to treat seizures, spasticity, dystonia and other neuropsychiatric conditions. The Sham intervention uses a sham magnetic coil.
  Other Names: rTMS, TBS, TMS
  Arms: Sham Repetitive Transcranial Magnetic Stimulation
Device: Active Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (RTMS) is a relatively new technology that allows for targeted noninvasive stimulation of the brain. RTMS is currently FDA-cleared for the treatment of refractory depression. It is also used experimentally to treat seizures, spasticity, dystonia and other neuropsychiatric conditions. The Active intervention uses an active magnetic coil.
  Other Names: rTMS, TBS, TMS
  Arms: Active Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Specific Aim1: Using a paradigm of Transcranial Magnetic Stimulation called Continuous Theta Burst Stimulation (cTBS) to reduce tics in Tourette Syndrome subjects

Hypothesis1: cTBS, compared to sham stimulation, will reduce tic severity by at least 25% as measured by the Yale Global Tic Severity Scale

Specific Aim2: Using cTBS to further understand neural correlates of tic generation

Hypothesis2: Functional MRI BOLD signal activation pattern will change after cTBS and this change will correlate with clinical improvement in tic severity

DETAILED DESCRIPTION:
Tourette syndrome (TS) is characterized by multiple motor and phonic tics. Current understanding of tic generation is thought involve the cortico-basal-thalamic-cortical circuit. At this time, only two medications are FDA-approved for tic treatment, while many more are used in an off-label fashion with only partial success. Despite multiple approaches for tic suppression, patients with severe tics are often left with inadequate relief. Repetitive Transcranial Magnetic Stimulation (RTMS) is a new technology which allows for noninvasive stimulation of the brain. In few pilot studies, RTMS reduced tic severity when targeting the Supplementary Motor Area (SMA). In this study, we propose to use a specific paradigm of RTMS called Continuous Theta Burst Stimulation (cTBS) over SMA to treat pediatric and adult patients with tics. We will utilize functional MRI (fMRI) to identify each subject's SMA for individualized stimulation. We hypothesize that this stimulation technique can reduce tic severity when compared to sham stimulation. This proposal is novel because 1) cTBS is offered as a new RTMS paradigm to reduce tics and 2) combination of RTMS and fMRI allows us to investigate the effects of cortical stimulation on the neural correlates of tic generation.

ELIGIBILITY:
Inclusion Criteria:1. Children or adults with Tourette Syndrome, tic disorder, chronic motor or vocal tics disorder ages 10 to 60 years.

2. Current tics with Yale Global Tic Severity Scale (YGTSS) score > 10. 3. If subject is on tic-suppressing medication(s) at the time of recruitment, no medication or dose changes allowed within the past seven days.

4. If subject receives botulinum toxin injection for tic management, the injection must be at least twelve weeks prior to the day of the study.

5. After the TBS sessions, no tic-suppression medications can be changed for at least one week.

6. All patients ages 10 to 60 years old with Tourette Syndrome, tic disorder, chronic motor or vocal tics disorder will be offered to participate in the study. If the patient decides to participate in the study, our study coordinator will obtain informed consent from the adult participant, or at least one parent of the pediatric participant. The consent form is written in English; the form is also written in a manner understandable by the person signing the form. The adult participant, the parent(s) of participant or the pediatric participant does not have to make a decision at the time of clinic visit, thus, minimizing coercion to participate.

-

Exclusion Criteria:1. Implanted brain stimulator, vagal nerve stimulator, VP shunt, aneurysm clip, cardiac pacemaker, or implanted medication port.

2. Prior ischemic or hemorrhagic stroke or traumatic brain injury. 3. History of seizure or epilepsy 4. If female, pregnant or sexually active and not using birth control. Abstinence will be permitted at the discretion of the TS clinicians, consistent with other IRB approved studies involving this population.

-

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Wu, MD, Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Repetitive Transcranial Magnetic Stimulation: In the active arm, patients received 8 sessions of active continuous theta burst stimulation (cTBS) over 2 consecutive days. Four 40-second cTBS sessions were given over a 75-minute period (0, 15, 60, 75 minute marks) for each day. We used Magstim 70mm figure-8 TMS coil, placed over SMA, with the coil handle pointing towards the occiput.
- Sham Repetitive Transcranial Magnetic Stimulation: In the sham arm, patients received 8 sessions of active continuous theta burst stimulation (cTBS) over 2 consecutive days. Four 40-second cTBS sessions were given over a 75-minute period (0, 15, 60, 75 minute marks) for each day. We used Magstim sham 70mm figure-8 TMS coil, placed over SMA, with the coil handle pointing towards the occiput.
Period: Overall Study
Arm/Group | Active Repetitive Transcranial Magnetic Stimulation | Sham Repetitive Transcranial Magnetic Stimulation
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Repetitive Transcranial Magnetic Stimulation | Sham Repetitive Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (3.9) | 15.5 (4) | 14.5 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 6 | 3 | 9
Yale Global Tic Severity Scale [Mean (Standard Deviation); unit: units on a scale (0 - 50)] — The tic severity score based on Yale Global Tic Severity Scale ranges from 0 - 50. A person who has no tics would have a score of 0. High score means a person has severe tics.
  units on a scale (0 - 50) | 27.5 (7.4) | 26.8 (4.8) | 27.2 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Scale
Description: The tic severity score based on Yale Global Tic Severity Scale ranges from 0 - 50. A person who has no tics would have a score of 0. High score means a person has severe tics.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale (0 - 50)
Arm/Group | Active Repetitive Transcranial Magnetic Stimulation | Sham Repetitive Transcranial Magnetic Stimulation
Number analyzed (Participants) | 6 | 6
units on a scale (0 - 50) | 23.2 (9.8) | 21.7 (7.7)

ADVERSE EVENTS:
Description: Systematic assessment for adverse events was performed using a 16-item Review of Systems.
Arm/Group | Active Repetitive Transcranial Magnetic Stimulation | Sham Repetitive Transcranial Magnetic Stimulation
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Repetitive Transcranial Magnetic Stimulation (N=6) | Sham Repetitive Transcranial Magnetic Stimulation (N=6)
Mild headache (Nervous system disorders) | 1 | 1
Mild abdominal discomfort (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No